CLINICAL TRIAL: NCT01689441
Title: Randomized Controlled Trial of Calcitriol vs. Placebo Among Critically-ill Patients With Sepsis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Leaf, Assistant Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012P001755
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Severe Sepsis or Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcitriol (Experimental): Calcitriol 2mcg IV x 1
  Interventions: Drug: Calcitriol
- Placebo (Placebo Comparator): Normal saline 2cc IV x 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitriol
  Arms: Calcitriol
Drug: Placebo
  Arms: Placebo

SUMMARY:
Observational studies among critically ill patients have shown strong associations between vitamin D deficiency and adverse outcomes, including increased length of stay, infection, and mortality. It is unknown whether vitamin D deficiency contributes directly to adverse outcomes or whether it is simply a biomarker of severity of illness or overall health status. However, vitamin D plays a key role in host defense, largely by stimulating production of the anti-microbial peptide cathelicidin (LL-37). We will test the hypothesis that administration of activated vitamin D (calcitriol) will increase serum levels of cathelicidin.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* Severe sepsis or septic shock
* Central venous catheter (for blood drawing)

Exclusion Criteria:

* Serum calcium ≥ 10.0 mg/dl or phosphate ≥ 6.0 mg/dl, assessed within previous 48 hours
* Current or recent therapy (within previous 7 days) with nutritional vitamin D at doses >1,000 I.U. per day or activated vitamin D at any dose
* History of solid organ or bone marrow transplant, primary parathyroid disease, metabolic bone disease, or sarcoidosis
* Expected to die or leave the ICU within 48 hours
* History of hypersensitivity or any allergic reaction to calcitriol
* End stage renal disease
* Acute Kidney Injury receiving intermittent renal replacement therapy
* Enrolled in a competing study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Leaf, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Leaf DE, Raed A, Donnino MW, Ginde AA, Waikar SS. Randomized controlled trial of calcitriol in severe sepsis. Am J Respir Crit Care Med. 2014 Sep 1;190(5):533-41. doi: 10.1164/rccm.201405-0988OC. PMID 25029202
- See also: Link to manuscript in pubmed — http://www.ncbi.nlm.nih.gov/pubmed/25029202

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcitriol: Calcitriol 2mcg IV x 1
  Calcitriol
- Placebo: Normal saline 2cc IV x 1
  Placebo
Period: Overall Study
Arm/Group | Calcitriol | Placebo
Started | 36 | 31
Completed | 36 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcitriol | Placebo | Total
Number analyzed (Participants) | 36 | 31 | 67
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [54 to 70] | 58 [49 to 69] | 64 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 22 | 15 | 37
Region of Enrollment [Number; unit: participants]
  United States | 36 | 31 | 67

OUTCOME MEASURES:

1. Primary Outcome: Plasma Cathelicidin (hCAP18) Protein Levels at 48 Hours
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 36 | 31
ng/ml | 76 [60 to 94] | 82 [70 to 100]
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Plasma Interleukin-6 (IL-6) Levels at 48 Hours
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 36 | 31
pg/ml | 41 [25 to 92] | 32 [21 to 85]
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; Test type: Superiority or Other; p = 0.51, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Urinary Neutrophil Gelatinase-associated Lipocalin (NGAL) / Creatinine Ratio at 48 Hours
Description: NGAL is a urinary marker of renal tubular injury. NGAL levels were normalized to the urinary creatinine concentration to account for the influence of dilution on biomarker concentrations.
Time Frame: 48 hours
Population: The discrepancy in "number of participants analyzed" for this outcome vs. other outcomes is due to urine samples not being available in all participants
Measure: Median (Inter-Quartile Range); unit: mg/mg
Arm/Group | Calcitriol | Placebo
Number analyzed (Participants) | 30 | 24
mg/mg | 0.6 [0.2 to 3.1] | 0.7 [0.3 to 2.7]
Statistical Analysis 1: Comparison: Calcitriol vs Placebo; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Calcitriol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/31
Other Adverse Events (participants affected / at risk) | 0/36 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No